CLINICAL TRIAL: NCT06586918
Title: Verification of a Perfusion Index Parameter in Adult Volunteers
Brief Title: Perfusion Index Parameter
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT23025OM2VLP
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-09

CONDITIONS: Perfusion; Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers

SUMMARY:
To evaluate the association between the Perfusion index parameter and an independent measure of perfusion.

DETAILED DESCRIPTION:
Perfusion index parameters measured with an Investigational Pulse Oximetry PCBA, paired with Market Released sensors, will be compared to perfusion levels measured by a FDA-cleared device equipped with a laser Doppler technology-based device for blood perfusion measurements. Continuous Perfusion index measurements will be taken during the test sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥18 years of age
2. Subject is able to participate for the duration of the study
3. Subject is willing to sign an informed consent
4. Subject weighs >40kg

Exclusion Criteria:

1. Previous injury or trauma to fingers or hands that may change blood flow or vascular supply and affect the ability to test sensors
2. Physiologic abnormalities that prevent proper application of pulse oximetry sensor
3. Severe contact allergies that cause a reaction to standard adhesive materials such as those found in medical sensors and electrodes.
4. Raynaud Syndrome
5. Repeated systolic blood pressure > 140mmHg -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Male or Female volunteers age ≥18 years, weighing greater than 40kgs.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Perfusion Index (PI) correlation to doppler measurement | 1 hour
  To confirm correlation of Perfusion Index measured by the investigational pulse oximeter PCBA and Market Released sensors to the laser doppler measure of skin perfusion (LDSP) as determined by an overall instantaneous (lag(0)) Spearman rank correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Randall M Clark, M.D., Principal Investigator — Medtronic Clinical Physiology Lab
Locations (1):
- Medtronic Clinical Physiology Lab, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No